CLINICAL TRIAL: NCT04847362
Title: Investigation of the Effect of Tele-Health Education Provided in the Postpartum Period in the Covid 19 Pandemic on the Depression, Attachment and Anxiety Levels of Women: A Randomized Controlled Study
Brief Title: The Effect of Tele-Health Education Provided in the Postpartum Period in the Covid 19 Pandemic
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, ASSOCIATE PROFESSOR, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11.04.2021-27076
Record Dates: First submitted 2021-04-12; First posted 2021-04-19 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Postpartum Depression; Anxiety State
Keywords: postpartum depression; mother-baby attachment; anxiety
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The mothers in this group will be given telehealth training for 4 weeks.
  Interventions: Behavioral: Experimental
- Control (No Intervention): Mothers in this group will not be given telehealth education, they will receive care within the scope of routine care.

INTERVENTIONS:
Behavioral: Experimental — education group
  Arms: Experimental

SUMMARY:
In the planned study, it was aimed to examine the effect of tele-education offered in the postpartum period in the covid 19 pandemic on the levels of depression, attachment and anxiety of women.

DETAILED DESCRIPTION:
In the planned study, it was aimed to examine the effect of tele-education offered in the postpartum period in the covid 19 pandemic on the levels of depression, attachment and anxiety of women.

ELIGIBILITY:
inclusion Criteria

* literate
* Giving birth at term (between 38-42 weeks of gestation)
* Being on the 7th Postpartum Day,
* Participation in the study is voluntary,
* Absence of any psychiatric illness,
* Women who have characteristics such as not using any psychiatric medication.
* Baby with normal birth weight and APGAR score of 8 and above
* Those who have not developed postpartum complications
* Speaks and understands Turkish

Exclusion Criteria:

women who do not meet the sample selection criteria

-

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2021-04-11 (Actual); Primary Completion 2021-11-22 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
postpartum depression | postpartum 6 weeks
  The Edinburgh Postnatal Depression Scale (EPDS) was used to detect depressive symptoms during the postpartum period [30]. EPDS is a 10-item questionnaire assessing the interviewee's depressive feelings from the seven days before the interview. The response of the questions is scored from 0-3, with higher scores indicating higher levels of depressive symptoms. The total EPDS score of a respondentcan range from 0 to 30.
postpartum depression | postpartum 3 months
  The Edinburgh Postnatal Depression Scale (EPDS) was used to detect depressive symptoms during the postpartum period [30]. EPDS is a 10-item questionnaire assessing the interviewee's depressive feelings from the seven days before the interview. The response of the questions is scored from 0-3, with higher scores indicating higher levels of depressive symptoms. The total EPDS score of a respondentcan range from 0 to 30.
postpartum mother-baby attachment | postpartum 6 weeks a
  Postpartum Attachment Scale: Early diagnosis of problems in mother-infant relationship Developed to provide and maternal filling4. The scale is a six-digit It has a Likert scale. Scale "always", Postpartum attachment scales in mothers 247 "Very often", "often", "sometimes", "rarely", "no It has been defined as "time". Items 0-5 It is rated as. Scale 17 is reverse It consists of 25 graded items. Scale "attachment disorder" (12 items), "Rejection and irritability" (seven items), "care tension about "(four items), abuse four sub-categories with risk (two substances) It consists of units. Pathology in mother-infant relationship cut point specified for four subscales 4'18 The cut-off point of four subscales attachment disorder (subscale 1), respectively> 12, rejection and irritability (subscale 2)> 17, anxiety in infant care (subscale 3)> 10, the risk of abuse (subscale 4) is> 3.
postpartum mother-baby attachment | postpartum 3 months
  Postpartum Attachment Scale: Early diagnosis of problems in mother-infant relationship Developed to provide and maternal filling4. The scale is a six-digit It has a Likert scale. Scale "always", Postpartum attachment scales in mothers 247 "Very often", "often", "sometimes", "rarely", "no It has been defined as "time". Items 0-5 It is rated as. Scale 17 is reverse It consists of 25 graded items. Scale "attachment disorder" (12 items), "Rejection and irritability" (seven items), "care tension about "(four items), abuse four sub-categories with risk (two substances) It consists of units. Pathology in mother-infant relationship cut point specified for four subscales 4'18 The cut-off point of four subscales attachment disorder (subscale 1), respectively> 12, rejection and irritability (subscale 2)> 17, anxiety in infant care (subscale 3)> 10, the risk of abuse (subscale 4) is> 3.
anxiety state | postpartum 6 weeks
  State Anxiety Scale (STAI-I) in 1970 Turkish form developed by Spielberger Oner N et al. Its validity and reliability study has been carried out by adapting it. Anxiety level In STAI-I, "(1) not at all, (2) a little, (3) a lot and (4) completely" While it is scored as, the options in STAI-II are (1) almost never, (2) sometimes, (3) a lot of time, and (4) it is almost always. 2 kinds of scales Scores obtained from both scales theoretically it ranges from 20 to 80. High score indicates high anxiety level
anxiety state | postpartum 3 months
  State Anxiety Scale (STAI-I) in 1970 Turkish form developed by Spielberger Oner N et al. Its validity and reliability study has been carried out by adapting it. Anxiety level In STAI-I, "(1) not at all, (2) a little, (3) a lot and (4) completely" While it is scored as, the options in STAI-II are (1) almost never, (2) sometimes, (3) a lot of time, and (4) it is almost always. 2 kinds of scales Scores obtained from both scales theoretically it ranges from 20 to 80. High score indicates high anxiety level

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Zeynep Kamil Women's and Children's Diseases Training and Research Hospital, Istanbul
  - Saglık Bilimleri Universitesi, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided